CLINICAL TRIAL: NCT03575832
Title: Watchful Living: A Lifestyle Intervention for Black and Hispanic Prostate Cancer Patients and Their Partners
Brief Title: Watchful Living in Improving Quality of Life in Participants With Localized Prostate Cancer on Active Surveillance and Their Partners
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2017-0556; NCI-2018-01406 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0556 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-06-20; First posted 2018-07-03 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Stage I Prostate Cancer AJCC v8; Stage II Prostate Cancer AJCC v8; Stage IIA Prostate Cancer AJCC v8; Stage IIB Prostate Cancer AJCC v8; Stage IIC Prostate Cancer AJCC v8; Stage III Prostate Cancer AJCC v8; Stage IIIA Prostate Cancer AJCC v8; Stage IIIB Prostate Cancer AJCC v8; Stage IIIC Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (exercise, nutrition counseling) (Experimental): Participants receive an exercise plan and printed materials at baseline. Participants also receive 10 telephone coaching calls over 45-60 minutes weekly during month 1, every 2 weeks during month 2, and every month during months 3-6. Participants complete 2 nutrition counseling sessions before month 3.
  Interventions: Other: Counseling; Other: Informational Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Behavioral: Telephone-Based Intervention

INTERVENTIONS:
Other: Counseling — Complete nutrition counseling sessions
  Other Names: Counseling Intervention
Other: Informational Intervention — Receive an exercise plan and printed materials
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Behavioral: Telephone-Based Intervention — Receive telephone coaching calls

SUMMARY:
This pilot trial studies how well Watchful Living works in improving quality of life in participants with prostate cancer that has not spread to other parts of the body who are on active surveillance and their partners. A social support lifestyle intervention (called Watchful Living) may help African American prostate cancer participants and their partners improve their quality of life, physical activity, diet, and inflammation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of recruiting and implementing a lifestyle intervention for prostate cancer patients and their partners.

SECONDARY OBJECTIVES:

I. To evaluate the preliminary efficacy of a lifestyle intervention in improving diet, physical activity, physical fitness, partner's support, quality of life, and inflammation at the end of the study (month 6).

II. To conduct a process evaluation of the lifestyle intervention. III. Explore participants' satisfaction, likes/dislikes, strengths, weaknesses, and areas of improvement regarding the program.

OUTLINE:

Participants receive an exercise plan and printed materials at baseline. Participants also receive 10 telephone coaching calls over 45-60 minutes weekly during month 1, every 2 weeks during month 2, and every month during months 3-6. Participants complete 2 nutrition counseling sessions before month 3.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as black or African American or Hispanic (patient)
* Be greater than 18 years of age (patient and spouse or intimate partner)
* Have 0-III stage prostate cancer (patient)
* If treated, have completed therapy (e.g., surgery, chemo and/or radiation) (patient)
* Enroll with a spouse or intimate partner (patient)
* Do not meet physical activity recommendation (i.e., 150 minutes of moderate intensity physical activity per week) (patient and spouse or intimate partner)
* Be ready and able to be physically active, as determined by a physician (letter from a physician or nurse practitioner) (patient and spouse or intimate partner)
* Not participate in another physical activity, diet, or lifestyle program (patient)
* Have a valid home address and telephone number (patient)
* Internet access at home or other location (e.g., work, church, library, community center, etc.) (spouse or intimate partner)
* Patients on active surveillance will be included

Exclusion Criteria:

* They have an active noncutaneous malignancy at any site (patient)
* Had prior radiation therapy for treatment of the primary tumor (patient)
* Have planned concomitant immunotherapy, hormonal therapy, chemotherapy, or radiation therapy during the study period (patient)
* Are enrolled in another active surveillance protocol (patient)
* Participated in formative focus groups for this study (patient and spouse or intimate partner)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment and retention | Up to 8 months
  Rates of study eligibility, recruitment, and retention will be assessed. Will maintain detailed information during the recruitment process regarding numbers of patients and their partners interested, eligible, ineligible (and reasons for ineligibility), and enrolled (and reasons for choosing not to enroll if deemed eligible). Will calculate rates of study eligibility, recruitment, and retention, along with 90% confidence intervals (CIs). Participant feedback will be summarized using means and standard deviations (SDs), along with graphical display (e.g., box plots). Will also assess reasons for withdrawal from study among those that chose to withdraw. Will examine the differences between dropout and non-dropout group at each time point by demographic factors such as age, gender, marital status, education, and income.
Intervention adherence | Up to 8 months
  The intervention adherence rate for each dyad is defined as the proportion of intervention sessions completed by both the patient and partner. Will also look at percentage of both patient and partner completing a minimum of 7 out of 10 coaching calls and both nutrition counseling sessions.

SECONDARY OUTCOMES:
Surveillance lifestyle | Up to 8 months
  Will report means, standard deviations, and distributions of survey measures (including pre-post changes of these measures, as appropriate) for ceiling/floor effects and restrictions in range. Outcome measures will be treated as continuous variables. Linear mixed models will be used when combined data from both patients and partners are analyzed due to their correlation within couples. Two-sided statistical tests will be performed, and the significance level for each test will be set at 0.05 without adjustment for multiple testing. All results from the statistical tests will be interpreted as hypothesis generating rather than conclusive findings. Will also perform paired t-tests to compare efficacy outcomes of interest between baseline and post intervention separately for patients and partners.
Elements of the intervention that were successful and/or need improvements | Up to 8 months
  Will conduct focus groups with a subsample of patient-partner dyads. Questions will address participants' experiences; thoughts about strengths, weaknesses, and needed improvements; perceptions about outcomes and impact; and overall reactions to and satisfaction with the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Lorna McNeill, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Harris Health System (LBJ), Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org